CLINICAL TRIAL: NCT02366351
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Clinical Trial to Evaluate the Pharmacokinetics/Pharmacodynamics, Efficacy and Safety of SHR3824 as Monotherapy in Chinese Subjects With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control
Brief Title: The PK/PD, Efficacy, Safety and Tolerability Study of SHR3824 in Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR3824-107
Record Dates: First submitted 2015-02-10; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — henagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- SHR3824 Placebo (Experimental): once daily, 12 weeks
  Interventions: Drug: Placebo
- SHR3824 5 mg (Experimental): once daily, 12 weeks
  Interventions: Drug: SHR3824
- SHR3824 10 mg (Experimental): once daily, 12 weeks
  Interventions: Drug: SHR3824
- SHR3824 20 mg (Experimental): once daily, 12 weeks
  Interventions: Drug: SHR3824

INTERVENTIONS:
Drug: SHR3824 — Once daily, 12 weeks
  Arms: SHR3824 10 mg; SHR3824 20 mg; SHR3824 5 mg
Drug: Placebo — Once daily, 12 weeks
  Arms: SHR3824 Placebo

SUMMARY:
The purpose of this study is to obtain information on PK/PD, efficacy and safety of SHR3824 over 12 weeks in Chinese patients with Type 2 Diabetes. This will be done by comparing the effect of SHR3824 to placebo when given in oral doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of type 2 diabetes mellitus;
* Hemoglobin A1c levels >=7.5% and <=10.5%;
* Body mass index (BMI) 25 to 45 kg/m2;
* Patient either has not been previously treated with antihyperglycemic medication or has not been treated with antihyperglycemic in the last 10 weeks.

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes mellitus (acromegaly, Cushing's syndrome, etc.);
* Past or current history of severe diabetic complications (proliferative diabetic retinopathy, stage III or later stage overt nephropathy, diabetic ketoacidosis, or serious diabetic neuropathy);
* Systolic blood pressure of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg on the start or end day of the run-in period;
* History of myocardial infarction, unstable angina, or cerebrovascular disorder within 6 months before the start of the run-in period;
* Past or current history of malignant tumor;
* Past or current history of drug hypersensitivity such as shock and anaphylactoid symptoms;
* Pregnant women, lactating mothers, or women of childbearing potential;
* Any condition that subjects are assessed to be ineligible by the investigator (sub investigator).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Adjusted Mean Change in HbA1c Levels | Baseline to Week 12
The number of volunteers with adverse events as a measure of safety and tolerability | Baseline to Week 12

SECONDARY OUTCOMES:
Adjusted Mean Change in Fasting Plasma Glucose | Baseline to Week 12
Proportion of Participants Achieving Glycemic Response Defined as HbA1c <7% | Baseline to Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China